CLINICAL TRIAL: NCT04441216
Title: Effects of a Novel Formulation of Traditional Chinese Medicine (TCM) For Prevention of Type 2 Diabetes (T2D)
Brief Title: Effects of TCM on Beta-cell Function and Insulin Resistance in High Risk Chinese Individuals for T2D (TCM_PDiab_P01)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Juliana Chan, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRE-2019.601
Record Dates: First submitted 2020-04-20; First posted 2020-06-22 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Prediabetic State
Keywords: Prediabetes; Chinese Medicine
MeSH Terms: conditions — Prediabetic State | interventions — Coptidis rhizoma extract; Huang Qi; lonicerae flos

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Consultation only (No Intervention): Review by Chinese Medicine practitioner only
- JinQi JiangTang Fang (Active Comparator): JinQi JiangTang Fang (Rhizoma Coptidis, Radix Astragali and Flos Lonicerae)
  Interventions: Other: Rhizoma Coptidis, Radix Astragali and Flos Lonicerae
- JM-ELD (Active Comparator): JQJT plus extra low dose Ophiopogonis Radix
  Interventions: Other: Rhizoma Coptidis, Radix Astragali and Flos Lonicerae, Ophiopogonis Radix
- JM-LD (Active Comparator): JQJT plus low doses Ophiopogonis Radix
  Interventions: Other: Rhizoma Coptidis, Radix Astragali and Flos Lonicerae, Ophiopogonis Radix

INTERVENTIONS:
Other: Rhizoma Coptidis, Radix Astragali and Flos Lonicerae — granule
  Arms: JinQi JiangTang Fang
Other: Rhizoma Coptidis, Radix Astragali and Flos Lonicerae, Ophiopogonis Radix — granule
  Arms: JM-ELD; JM-LD

SUMMARY:
This study involves prediabetes volunteers who are at high risk of developing diabetes, including those with family history of diabetes, metabolic syndrome, fatty liver, polycystic ovary syndrome and history of gestational diabetes. They will take a 12-week course of formula: a) JinQi JiangTang Fang (JQJT) including Coptidis Rhizoma, Astragali Radix and Lonicerae Japonicae Flos, b) combined the ingredients of JQJT and Ophiopogonis Radix to make up a novel CM, Jin Mai Fang (JM); to evaluate the effectiveness of Chinese Medicine in preventing diabetes in a controlled setting in order to better understand their actions. They will be followed up for another 12 weeks after the treatment to evaluate the improvement in glucose tolerance of the formula.

DETAILED DESCRIPTION:
In China, 10% of adults have diabetes and 30% of people have prediabetes. In Hong Kong, 2 in 100 adults develop pre-diabetes every year and in 2014, 9% of adults have prediabetes. People with prediabetes have increased risk of cardiovascular disease and development of diabetes. Once developed, diabetes is associated with loss of 4-10 years of life depending on age of onset and 2-3 fold increased risk of cardiovascular, kidney and cancer events.

Early detection and intervention of pre-diabetes will prevent progression from pre-diabetes to diabetes and reduce the risk of complications of diabetes. This focus on prevention concords with the concept of 'Zhi-Wei-Bing' in Chinese Medicine (CM). This is not only an important philosophy of CM but also a unique feature of Chinese culture. The 'Zhi-Wei-Bing' philosophy includes disease prevention, treatment, and rehabilitation.

Insulin is secreted by the beta-cells of the pancreas which is the only hormone that can reduce blood glucose. People with diabetes have fewer pancreatic beta-cells than those without diabetes. Chinese Medicine contains multiple herbs which have been used in China for thousands of years. These herbal mixtures may alter the expression of these proteins which can lead to many biological effects including the possible benefits in reducing the risk of diabetes in high risk subjects.

JinQi JiangTang Fang (JQJT) contains extracts from three herbs including Coptidis Rhizoma, Astragali Radix and Lonicerae Japonicae Flos and is one of the most popular formulae used by CMP for prevention of diabetes. The sustained blood glucose lowering effects of JQJT in male Zucker diabetic fatty rats. On multiomic analysis, the investigators observed concerted expression changes in a gene-gene network involving mRNA, miRNA and proteins implicated in fat metabolism and cell cycles.

In this study, the investigators have combined the ingredients of JQJT and Ophiopogonis Radix (Maidong) to make up a novel CM formula, Jin Mai Fang (JM). According to TCM theory, Maidong nourishes the yin, promotes body fluid production, moistens the lung, eases the mind and clears away heart fire. The polysaccharide-rich extract of Maidong (0.06-240 mg/ml) has been shown to inhibit glucose absorption into the intestinal brush border membrane vesicles, reduce the activity of α-glucosidase and improve the activity of NIT-1 cells damaged by streptozotocin. These combined effects of inhibition of carbohydrate digestion and absorption and protection of the pancreatic islet cells provide a strong rationale for its use to prevent diabetes. The subjects will take a 12-week course of formula and they will be followed up for another 12 weeks after the treatment to evaluate the improvement in glucose tolerance of the formula.

ELIGIBILITY:
Inclusion criteria

* Individuals aged ≥18 years-70 years
* BMI≥18 kg/m2
* Chinese ethnicity
* Individuals with pre-diabetes based on 75 gram oral glucose tolerance test (OGTT) defined as impaired fasting glycemia (fasting plasma glucose (FPG): ≥5.6-6.9 mmol/L) and/or impaired glucose tolerance (IGT) (2-h PG: ≥7.8-11.0 mmol/L) -
* Plus at least one risk factor(s) from the following list:
* 2 components of the metabolic syndrome

  * Triglyceride≥1.7 mmol/L
  * BP≥130/80 mmHg
  * HDL-C<1.3 mmol/L in women or <1.1 mmol/L in men
  * Waist circumference≥80 cm in women or ≥90 cm in men
* Fatty liver

  * Diagnosis by ultrasound scan and/or
  * Diagnosis by fibroscan and/or
  * Diagnosis by ALT>35 IU/L in men and >24 IU/L in women
* History of diabetes in first degree relatives
* History of gestational diabetes mellitus
* History of polycystic ovary syndrome

Exclusion criteria

* Not willing to participate in this study or adhere to study procedures
* Significant medical history including but not limited to history of CVD, renal estimated glomerular filtration rate (eGFR) <60 ml/min/1.73m2 and/or liver dysfunction (AST and/or ALT≥3 times upper limit of normal)
* History of drug abuse or excessive alcohol intake based on investigator judgment
* Dehydration, diarrhea or vomiting at the time of recruitment
* Subjects with severe infection, in perioperative period or with serious injury at the time of recruitment
* Subjects with blood haemoglobin outside the normal range (male: 13.5-17.5 g/dl and female: 12-15.5 g/dl)
* Subjects who have donated blood in the 3 months prior to the study and/or plan to donate blood during the study period
* Current use of dietary supplements or health products affecting glycose or galactose metabolism or body weight in previous 1 month before first dosing.
* Breast feeding, pregnant women or women with plans for pregnancy
* Any conditions considered unsuitable by the investigators
* Subjects with use of Warfarin
* Subjects with known G6PD deficiency or known history of herb-drug interactions
* Known history of diabetes mellitus and/or HbA1c >= 6.5%.
* Usage of glucose lowering drugs and/or weight loss drugs currently or within 1 month before first dosing
* Previous metabolic surgery
* Known history of thyroid disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-02 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Between-group differences in glycemic excursion during 75g OGTT as indicated by area under the curve (AUC) plasma glucose concentration during 12-week on-treatment and 12-week off treatment period | 24 weeks
  Plasma glucose during 75g OGTT will be measured at baseline, after 12 weeks treatment and 12 weeks of treatment period

SECONDARY OUTCOMES:
Between group differences in insulin resistance (HOMA-IR),as indicated by area under the curve (AUC) plasma insulin during 12-week on-treatment and 12-week off treatment period | 24 weeks
  Plasma insulin during 75g OGTT will be measured at baseline, after 12 weeks treatment and 12 weeks of treatment period
Between group differences in beta-cell function (HOMA-beta) as indicated by area under the curve (AUC) plasma insulin during 12-week on-treatment and 12-week off treatment period | 24 weeks
  Plasma insulin during 75g OGTT will be measured at baseline, after 12 weeks treatment and 12 weeks of treatment period
Between group differences in quantitative insulin sensitivity check index (QUICKI) as indicated by during 12-week on-treatment and 12-week off treatment period | 24 weeks
  Plasma insulin during 75g OGTT will be measured at baseline, after 12 weeks treatment and 12 weeks of treatment period
Between group differences in insulinogenic index as indicated by during 12-week on-treatment and 12-week off treatment period | 24 weeks
  Plasma insulin during 75g OGTT will be measured at baseline, after 12 weeks treatment and 12 weeks of treatment period
Between group differences in vital sign during 12-week on-treatment and 12-week off treatment period | 24 weeks
  Measure blood pressure at baseline, after 12 weeks treatment and 12 weeks of treatment period
Between group differences in body weight during 12-week on-treatment and 12-week off treatment period | 24 weeks
  Measure body weight at baseline, after 12 weeks treatment and 12 weeks of treatment period
Between group differences in renal function during 12-week on-treatment and 12-week off treatment period | 24 weeks
  Measure renal function test by measuring Serum creatinine test at baseline, after 12 weeks treatment and 12 weeks of treatment period
Between group differences in liver function during 12-week on-treatment and 12-week off treatment period | 24 weeks
  Measure liver function test by measuring the change of Alanine transaminase (ALT) test at baseline, after 12 weeks treatment and 12 weeks of treatment period
Prevalence of euglycaemic chinese subject after 12-week on-treatment and 12-week off treatment period | 24 weeks
  investigate the proportion of reversal from pre-diabetes to euglycaemia by assessing number euglycaemic subject after 12 weeks on treatment and 12 weeks off treatment period

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong